CLINICAL TRIAL: NCT03934060
Title: Effects of a Specific Strength Training Regarding Activities of Daily Living (ADLs) Associated With Movement During Treatment of Leukemia or Non-Hodgkin Lymphoma in Childhood and Adolescence
Brief Title: Strength Training and ADLs in Childhood Leukemia and Lymphoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Sabine Kesting, Prinzipal Investigator, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DJCLS 15 R/2016
Record Dates: First submitted 2019-04-14; First posted 2019-05-01 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Childhood Cancer
Keywords: exercise; strength training; activities of daily living; childhood cancer; leukemia; Non-Hodgkin lymphoma
MeSH Terms: conditions — Neoplasms; Motor Activity; Leukemia; Lymphoma, Non-Hodgkin | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Supervised exercise training including specific strength training tools and general exercise contents (standard care), 2-3 times per week, 30 minutes per session
  Interventions: Other: Exercise
- Control (No Intervention): Supervised exercise training regarding general exercise contents (standard care), 2-3 times per week, 30 min per session

INTERVENTIONS:
Other: Exercise — specific strength training
  Arms: Intervention

SUMMARY:
Reduced activity levels and reduced muscular strength could severely impair the activities of daily living (ADLs) in pediatric leukemia and Non-Hodgkin lymphoma patients. Increased muscle strength is associated with improved accomplishment of ADLs and consequently greatest possible normality, autonomy and mobility. Primary outcome of this RCT (n=20/20) is the analysis of effects of a treatment-associated and close to every day life strength training (2-3 times/week) compared to a general exercise program (standard care).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Acute Leukemia or Non-Hodgkin Lymphoma
* Diagnosed and/or treated at the Kinderklinik München Schwabing, Technische Universität München
* Informed consent as documented by signature

Exclusion Criteria:

* Medical contraindications regarding strength training (e.g. risk of bleeding, ...)
* Contraindications to one of the inclusion criteria mentioned above
* Inability to follow the procedures and understand the intervention and assessments of this study, e.g. due to cognitive impairment, language problems, psychological disorders etc.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Change of score of the Activities Scale for Kids - performance version | Change of the ASK score from baseline to 3 months, change from 3 months to 6 months, change from 6 months to 12 months
  The ASK - Activities Scale for Kids performance version by NL Young assesses an overall summary score (0-100) of self-reported activities of daily living in children and adolescents. The scale monitors changes associated with therapeutic interventions. Higher values represent a better outcome. The ASK contains 30 items in 7 sub-domains (personal care, dressing, other skills, locomotion, play, standing skills and transfer).

SECONDARY OUTCOMES:
Change of motor performance analyzed with the Motor performance test in Pediatiric Oncology (MOON) | Change of motor performance from baseline to 6 months
  Motor performance is assessed by the MOON-test, a tool to examine motor performance abilities in children and adolescents during and after cancer treatment. There's no summary score; reference values of healthy children enable comparison of the tested children.
Change of level of physical activity | Change of physical activity level from baseline to 3 months, from 3 to 6 months, from 6 to 12 months
  Physical activity is assessed using an accelerometer (movisens) for the period of 7 days.
Change in performance in a parkour in activities of daily living | Change of score in the parkour from baseline to 6 months
  A standardized parkour with tasks imitating activities of daily living is used to objectively verify the ASK score. Points from 0-4 are counted for each task depending on quality of movement (0 = task can not be completed, 1 = task can be completed with help, 2 = task can be completed with several attempts, 3 = task can be completed with only little effort, 4 = task can be completed without any problems or effort). There are no reference values for the parkour, but intra-individual changes are analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Kinderklinik München Schwabing TUM School of Medicine, Department of Pediatrics and Children's Cancer Research Center, Technical University of Munich, Munich, Bavaria, Germany